CLINICAL TRIAL: NCT03556358
Title: A Randomized, Double-blind, Parallel Group, Phase III Trial to Compare the Efficacy, Safety, and Immunogenicity of TX05 With Herceptin® in Subjects With HER2 Positive Early Breast Cancer
Brief Title: Trial to Compare the Safety, Efficacy and Immunogenicity of TX05 With Herceptin® in HER2+ Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanvex BioPharma USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TX05-03
Record Dates: First submitted 2018-06-01; First posted 2018-06-14 (Actual); Results first posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Breast Neoplasms; HER2-positive Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
Keywords: trastuzumab; Herceptin
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TX05 (trastuzumab) (Experimental): • Intravenous (IV) epirubicin, 75 mg/m^2 and cyclophosphamide 600 mg/m2 every 3 weeks for 4 cycles
  Followed by:
  • IV TX05 8 mg/kg loading dose then 6 mg/kg and paclitaxel 175 mg/m2 every 3 weeks for 4 cycles
  Interventions: Biological: TX05 (trastuzumab); Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide
- Herceptin® (Active Comparator): • Intravenous (IV) epirubicin, 75 mg/m^2 and cyclophosphamide 600 mg/m2 every 3 weeks for 4 cycles
  Followed by:
  • IV Herceptin 8 mg/kg loading dose then 6 mg/kg and paclitaxel 175 mg/m2 every 3 weeks for 4 cycles
  Interventions: Biological: Herceptin®; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: TX05 (trastuzumab) — 8 mg/kg, 90 min IV infusion (Cycle 5), followed by 6 mg/kg, 60 min IV infusion (Cycles 6 - 8)
  Arms: TX05 (trastuzumab)
Biological: Herceptin® — 8 mg/kg, 90 min IV infusion (Cycle 5), followed by 6 mg/kg, 60 min IV infusion (Cycles 6 - 8)
  Arms: Herceptin®
Drug: Paclitaxel — 175 mg/m^2, 60 min IV infusion, every 3 weeks (Cycles 5-8)
  Other Names: Ribotax
Drug: Epirubicin — 75 mg/m^2, IV bolus infusion, every 3 weeks (Cycles 1-4)
Drug: Cyclophosphamide — 600 mg/m^2, 30 min IV infusion, every 3 weeks (Cycles 1-4)

SUMMARY:
This is a Phase III, double-blind, randomized, multicenter study to compare the efficacy and to evaluate the safety and immunogenicity of TX05 (trastuzumab) with Herceptin® in subjects with HER2 positive early breast cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed HER 2 overexpressing invasive primary operable Stage II/IIIa breast cancer (AJCC version 7 staging criteria).
* Available tumor tissue for central review of HER2 status.
* Planned surgical resection of breast tumor.
* Planned neoadjuvant chemotherapy.
* Documentation of HER2 gene amplification or overexpression.
* Ipsilateral, measurable tumor longest diameter > 2 cm.
* Known estrogen receptor (ER) and progesterone receptor (PR) hormone status (may be performed during screening).
* ECOG performance status of 0 or 1.
* Adequate bone marrow, hepatic and renal functions.
* Left ventricular ejection fraction (LVEF) ≥ 50% or within institutional normal limits, measured by echocardiography or MUGA scan.
* Effective contraception as defined by protocol.

Key Exclusion Criteria:

* Investigational therapy within 2 months of first dose of study drug.
* Bilateral breast cancer.
* Inflammatory breast cancer
* Metastases.
* Prior chemotherapy, biologic therapy, radiation or surgery for any active malignancy, including breast cancer.
* Cardiac insufficiency, myocardial infarction, coronary/peripheral artery bypass graft, congestive heart failure, cerebrovascular accident, unstable angina pectoris, uncontrolled arrhythmia or pulmonary embolus within the previous 12 months prior to 1st administration of study drug.
* Clinically significant active infection, poorly controlled diabetes mellitus and/or uncontrolled hypertension.
* Major surgery, significant traumatic injury, radiation therapy and/or grade 3 hemorrhage within 4 weeks of 1st administration of study drug.
* Pre-existing clinically significant Grade 2 peripheral neuropathy.
* Malignancy within the last 5 years (except squamous/basal cell carcinoma of the skin, cervical carcinoma in situ and superficial bladder cancer).
* Severe dyspnea at rest requiring oxygen therapy.
* Known positive HIV, acute or chronic active infection with Hepatitis B or Hepatitis C.
* Current pregnancy or breastfeeding.
* Pre-existing thyroid abnormality with thyroid function that cannot be maintained in normal range despite optimal therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 809 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Mills, PhD, Study Director — Tanvex BioPharma USA, Inc.
Locations (146):
- Belarus (7):
  - Tanvex Investigational Site 1008, Lyasny, Minsk Oblast
  - Tanvex Investigational Site 1007, Babruysk, Mogilyov Oblast
  - Tanvex Investigational Site 1006, Grodno
  - Tanvex Investigational Site 1003, Homyel
  - Tanvex Investigational Site 1002, Minsk
  - Tanvex Investigational Site 1005, Mogilev
  - Tanvex Investigational Site 1001, Vitebsk
- Chile (2):
  - Tanvex Investigational Site 4001, Temuco
  - Tanvex Investigational Site 4002, Viña del Mar
- Georgia (13):
  - Tanvex Investigational Site 5006, Batumi
  - Tanvex Investigational Site 5002, Batumi
  - Tanvex Investigational Site 5003, Tbilisi
  - Tanvex Investigational Site 5001, Tbilisi
  - Tanvex Investigational Site 5005, Tbilisi
  - Tanvex Investigational Site 5012, Tbilisi
  - Tanvex Investigational Site 5013, Tbilisi
  - Tanvex Investigational Site 5004, Tbilisi
  - Tanvex Investigational Site 5010, Tbilisi
  - Tanvex Investigational Site 5011, Tbilisi
  - Tanvex Investigational Site 5008, Tbilisi
  - Tanvex Investigational Site 5009, Tbilisi
  - Tanvex Investigational Site 5007, Tbilisi
- Hungary (6):
  - Tanvex Investigational Site 6003, Budapest
  - Tanvex Investigational Site 6007, Budapest
  - Tanvex Investigational Site 6005, Debrecen
  - Tanvex Investigational Site 6006, Győr
  - Tanvex Investigational Site 6004, Miskolc
  - Tanvex Investigational Site 6001, Pécs
- India (27):
  - Tanvex Investigational Site 7007, Nashik, Maharashtra
  - Tanvex Investigational Site 7015, Pune, Maharashtra
  - Tanvex Investigational Site 7003, Pune, Maharashtra
  - Tanvex Investigational Site 7004, Pune, Maharashtra
  - Tanvex Investigational Site 7002, Bikaner, Rajasthan
  - Tanvex Investigational Site 7010, Madurai, Tamil Nadu
  - Tanvex Invesitgational Site 7033, Ahmedabad
  - Tanvex Investigational Site 7019, Bangalore
  - Tanvex Investigational Site 7037, Bangalore
  - Tanvex Investigational Site 7022, Belagavi
  - Tanvex Investigational Site 7034, Chandigarh
  - Tanvex Investigational Site 7013, Coimbatore
  - Tanvex Investigational Site 7024, Gūrgaon
  - Tanvex Investigational Site 7045, Hyderabad
  - Tanvex Investigational Site 7036, Hyderabad
  - Tanvex Investigational Site 7009, Jaipur
  - Tanvex Investigational Site 7039, Kolkata
  - Tanvex Investigational Site 7040, Kolkata
  - Tanvex Investigational Site 7006, Kolkata
  - Tanvex Investigational Site 7005, Lucknow
  - Tanvex Investigational Site 7012, Manipal
  - Tanvex Investigational Site 7041, Model Town
  - Tanvex Investigational Site 7001, Nashik
  - Tanvex Investigational Site 7031, Nāka
  - Tanvex Investigational Site 7042, Trichy
  - Tanvex Investigational Site 7018, Vadodara
  - Tanvex Investigational Site 7017, Vijayawada
- Mexico (14):
  - Tanvex Investigational Site 2102, Monterrey, Nuevo León
  - Tanvex Investigational Site 2117, Aguascalientes
  - Tanvex Investigational Site 2109, Aguascalientes
  - Tanvex Investigational Site 2116, Cancún
  - Tanvex Investigational Site 2104, Cuauhtémoc
  - Tanvex Investigational Site 2114, Cuauhtémoc
  - Tanvex Investigational Site 2101, Cuautitlán Izcalli
  - Tanvex Investigational Site 2111, Mexico City
  - Tanvex Investigational Site 2113, México
  - Tanvex Investigational Site 2103, Monterrey
  - Tanvex Investigational Site 2106, Oaxaca City
  - Tanvex Investigational Site 2112, San Luis Potosí City
  - Tanvex Investigational Site 2110, Tequisquiapan
  - Tanvex Investigational Site 2108, Zapopan
- Peru (11):
  - Tanvex Investigational Site 1104, Chiclayo, Lambayeque
  - Tanvex Investigational Site 1112, Lima Cercado, Lima region
  - Tanvex Investigational Site 1108, San Borja, Lima region
  - Tanvex Investigational Site 1113, San Borja, Lima region
  - Tanvex Investigational Site 1101, Arequipa
  - Tanvex Investigational Site 1107, Arequipa
  - Tanvex Investigational Site 1110, Lima
  - Tanvex Investigational Site 1105, San Isidro
  - Tanvex Investigational Site 1102, San Isidro
  - Tanvex Investigational Site 1109, Surquillo
  - Tanvex Investigational Site 1103, Trujillo
- Philippines (12):
  - Tanvex Investigational Site 1210, Santo Tomas, Batangas
  - Tanvex Investigational Site 1203, Cebu City, Cebu
  - Tanvex Investigational Site 1204, Cebu City, Cebu
  - Tanvex Investigational Site 1211, Cebu City, Cebu
  - Tanvex Investigational Site 1208, Quezon City, Manila
  - Tanvex Investigational Site 1207, Manila, National Capital Region
  - Tanvex Investigational Site 1206, Bacolod City, Negros Occidental
  - Tanvex Investigational Site 1212, Davao City
  - Tanvex Investigational Site 1214, Makati City
  - Tanvex Investigational Site 1201, Manila
  - Tanvex Investigational Site 1209, Quezon City
  - Tanvex Investigational Site 1213, Quezon City
- Russia (35):
  - Tanvex Investigational Site 1522, Ufa, Bashkortostan Republic
  - Tanvex Investigational Site 1529, Krasnodar, Krasnodarskiy Kray
  - Tanvex Investigational Site 1513, Sochi, Krasnodarskiy Kray
  - Tanvex Investigational Site 1509, Omsk, Omsk Oblast
  - Tanvex Investigational Site 1510, Pushkin, Sankt-Peterburg
  - Tanvex Investigational Site 1511, Novosibirsk, Siberia
  - Tanvex Investigational Site 1519, Pyatigorsk, Stavropol Kray
  - Tanvex Investigational Site 1518, Tomsk, Tomsk Oblast
  - Tanvex Investigational Site 1535, Arkhangelsk
  - Tanvex Investigational Site 1531, Belgorod
  - Tanvex Investigational Site 1538, Chelyabinsk
  - Tanvex Investigational Site 1520, Ivanovo
  - Tanvex Investigational Site 1515, Izhevsk
  - Tanvex Investigational Site 1502, Kaluga
  - Tanvex Investigational Site 1540, Kazan'
  - Tanvex Investigational Site 1512, Krasnoyarsk
  - Tanvex Investigational Site 1505, Kursk
  - Tanvex Investigational Site 1530, Moscow
  - Tanvex Investigational Site 1536, Moscow
  - Tanvex Investigational Site 1514, Moscow
  - Tanvex Investigational Site 1507, Moscow
  - Tanvex Investigational Site 1503, Omsk
  - Tanvex Investigational Site 1537, Orenburg
  - Tanvex Investigational Site 1521, Rostov-on-Don
  - Tanvex Investigational Site 1516, Saint Petersburg
  - Tanvex Investigational Site 1517, Saint Petersburg
  - Tanvex Investigational Site 1523, Saint Petersburg
  - Tanvex Investigational Site 1524, Saint Petersburg
  - Tanvex Investigational Site 1525, Saint Petersburg
  - Tanvex Investigational Site 1506, Saint Petersburg
  - Tanvex Investigational Site 1526, Saint Petersburg
  - Tanvex Investigational Site 1501, Saint Petersburg
  - Tanvex Investigational Site 1508, Saransk
  - Tanvex Investigational Site 1533, Tomsk
  - Tanvex Investigational Site 1534, Yaroslavl
- Ukraine (19):
  - Tanvex Investigational Site 1808, Chernihiv
  - Tanvex Investigational Site 1821, Chernivtsi
  - Tanvex Investigational Site 1803, Dnipro
  - Tanvex Investigational Site 1824, Dnipro
  - Tanvex Investigational Site 1820, Kherson
  - Tanvex Investigational Site 1812, Khmelnytskyi
  - Tanvex Investigational Site 1815, Kiev
  - Tanvex Investigational Site 1811, Kiev
  - Tanvex Investigational Site 1802, Kiev
  - Tanvex Investigational Site 1814, Kropyvnytskyi
  - Tanvex Investigational Site 1819, Kropyvnytskyi
  - Tanvex Investigational Site 1804, Kryvyi Rih
  - Tanvex Investigational Site 1809, Kyiv
  - Tanvex Investigational Site 1810, Odesa
  - Tanvex Investigational Site 1806, Sumy
  - Tanvex Investigational Site 1822, Ternopil
  - Tanvex Investigational Site 1823, Uzhhorod
  - Tanvex Investigational Site 1818, Vinnitsya
  - Tanvex Investigational Site 1813, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 809 subjects were randomized to the study. Of these, 806 subjects initiated protocol treatment.
Pre-assignment Details: Of the 806 subjects who initiated protocol treatment, 794 subjects initiated Cycle 5 (when trastuzumab was added); of these 394 subjects received TX05 and 400 subjects received Herceptin.
Groups:
- TX05 (Trastuzumab): • Intravenous (IV) epirubicin, 75 mg/m^2 and cyclophosphamide 600 mg/m2 every 3 weeks for 4 cycles
  Followed by:
  • IV TX05 8 mg/kg loading dose then 6 mg/kg and paclitaxel 175 mg/m2 every 3 weeks for 4 cycles
  TX05 (trastuzumab): 8 mg/kg, 90 min IV infusion (Cycle 5), followed by 6 mg/kg, 60 min IV infusion (Cycles 6 - 8)
  Paclitaxel: 175 mg/m^2, 60 min IV infusion, every 3 weeks (Cycles 5-8)
  Epirubicin: 75 mg/m^2, IV bolus infusion, every 3 weeks (Cycles 1-4)
  Cyclophosphamide: 600 mg/m^2, 30 min IV infusion, every 3 weeks (Cycles 1-4)
- Herceptin®: • Intravenous (IV) epirubicin, 75 mg/m^2 and cyclophosphamide 600 mg/m2 every 3 weeks for 4 cycles
  Followed by:
  • IV Herceptin 8 mg/kg loading dose then 6 mg/kg and paclitaxel 175 mg/m2 every 3 weeks for 4 cycles
  Herceptin®: 8 mg/kg, 90 min IV infusion (Cycle 5), followed by 6 mg/kg, 60 min IV infusion (Cycles 6 - 8)
  Paclitaxel: 175 mg/m^2, 60 min IV infusion, every 3 weeks (Cycles 5-8)
  Epirubicin: 75 mg/m^2, IV bolus infusion, every 3 weeks (Cycles 1-4)
  Cyclophosphamide: 600 mg/m^2, 30 min IV infusion, every 3 weeks (Cycles 1-4)
Period: Overall Study
Arm/Group | TX05 (Trastuzumab) | Herceptin®
Started | 404 | 405
Subjects Treated (Treated: Subjects treated with epirubicin and /or cyclophosphamide in cycle 1.) | 401 | 405
Subjects Receiving TX05 or Herceptin (TX05 or Herceptin was received at Cycle 5) | 394 | 400
Completed | 393 | 393
Not Completed | 11 | 12
Not completed — Subjects Randomized that did not Treat | 3 | 0
Not completed — Subjects who Randomized and Treated but Drop prior to Cycle 5 | 7 | 5
Not completed — Discontinued Treatment after Cycle 5 due to Adverse Event | 0 | 1
Not completed — Discontinued Treatment after Cycle 5 due to Death | 0 | 1
Not completed — Discontinued Treatment after Cycle 5 due to Consent Withdrawn | 0 | 2
Not completed — Discontinued Treatment after Cycle 5 due to COVID-19 | 0 | 1
Not completed — Discontinued Treatment after Cycle 5 due to Other (Subject Decision) | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety population/The modified intent-to-treat (mITT) population includes all subjects who are randomized into the study and receive at least 1 dose of TX05 or Herceptin.
Groups:
- Total: Total of all reporting groups
Arm/Group | TX05 (Trastuzumab) | Herceptin® | Total
Number analyzed (Participants) | 394 | 400 | 794
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (11.80) | 53.4 (10.83) | 53.8 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 394 | 400 | 794
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 71 | 140
  Not Hispanic or Latino | 325 | 328 | 653
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 14 | 29
  Asian | 64 | 72 | 136
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 292 | 286 | 578
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 23 | 27 | 50
Hormone Receptor Status [Count of Participants; unit: Participants]
  Positive | 253 | 254 | 507
  Negative | 141 | 146 | 287
ECOG [Count of Participants; unit: Participants] — Grade 0: Fully active, able to carry on all pre-disease activities without restriction
  Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  Grade 2: Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Grade 3: Capable of only limited self-care, confined to bed or chair more than 50% of waking hours.
  Grade 4: Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair.
  Grade 5: Dead
  Participants
    Grade 0 | 316 | 305 | 621
    Grade 1 | 78 | 95 | 173
Tumor Stage [Count of Participants; unit: Participants] — * Enrolled subjects should have Stage II/IIIa breast cancer.
  * Stage will be determined by the American Joint Committee on Cancer (AJCC) TNM (tumor size, lymph node involvement, metastasis to distant sites) staging system.
  * A low grade number (grade 1) usually means the cancer is slower-growing and less likely to spread. A high grade number (grade 3) means a faster-growing cancer that's more likely to spread. An intermediate grade number (grade 2) means the cancer is growing faster than a grade 1 cancer but slower than a grade 3 cancer.
  Participants
    IIA | 142 | 141 | 283
    IIB | 169 | 173 | 342
    IIIA | 83 | 86 | 169

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Each Treatment Arm Who Achieve Pathologic Complete Response (pCR)
Description: Pathologic complete response was determined by central review and defined as the absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled lymph nodes following neoadjuvant systemic therapy (ypT0/Tis ypN0).
Time Frame: 3-7 weeks following last dose of study treatment
Population: Per Protocol Population [includes all subjects who received at least one dose of study drug (TX05 or Herceptin) and had no major protocol deviations that impact the efficacy endpoints].
Measure: Number; unit: participants
Arm/Group | TX05 (Trastuzumab) | Herceptin®
Number analyzed (Participants) | 336 | 338
participants
  Subjects who do not Meet pCR Criteria | 172 | 185
  Subjects Meeting pCR Criteria | 164 | 153
Statistical Analysis 1: Comparison: TX05 (Trastuzumab) vs Herceptin®; Test type: Equivalence — Two one-sided hypothesis tests were performed for pCR in order to show that TX05 is equivalent to Herceptin: * TEST 1: H0a: θ1 / θ2 > 1.325 vs. H1a: θ1 / θ2 < 1.325 * TEST 2: H0b: θ1 / θ2 < 0.755 vs. H1b: θ1 / θ2 > 0.755 Where θ1 is the proportion of pCR for subjects randomized to TX05 group, θ2 is the proportion of pCR for subjects randomized to Herceptin. Equivalence was concluded if the 95% CI of the risk ratio is completely contained within the pre-defined interval [0.755, 1.325]; Risk Ratio (RR) = 1.0783, 95% CI 2-sided [0.9185 to 1.2659]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (ORR) = CR + PR.
Time Frame: End of Treatment (Week 24) or Early Termination Visit
Population: This analysis was performed on the modified intent-to-treat population. The modified intent-to-treat (mITT) population includes all subjects who were randomized and received at least 1 dose of TX05 or Herceptin.
Measure: Count of Participants; unit: Participants
Arm/Group | TX05 (Trastuzumab) | Herceptin®
Number analyzed (Participants) | 394 | 400
Participants | 332 | 340

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were recorded from Screening, while Adverse Events were recorded from Day 1 (Week 0) of Cycle 1 of study treatment through End of Treatment (Week 24).
Description: Because study drug (TX05/trastuzumab) was not introduced until Cycle 5 of treatment, the analyses of AEs was focused on Cycles 5 through 8 of treatment. The following results include events that occurred on or after initiation of TX05 or Herceptin treatment.
Arm/Group | TX05 (Trastuzumab) | Herceptin®
All-Cause Mortality (participants affected / at risk) | 0/394 | 1/400
Serious Adverse Events (participants affected / at risk) | 11/394 | 9/400
Other Adverse Events (participants affected / at risk) | 246/394 | 250/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TX05 (Trastuzumab) (N=394) | Herceptin® (N=400)
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 | 0
Vaginal Hemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2
Gastrointestinal Inflammation (Gastrointestinal disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Anaphylactic Reaction (Immune system disorders) | 0 | 1
Post Procedural Hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ischemic Stroke (Nervous system disorders) | 0 | 1
Fetal Death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0
COVID-19 Pneumonia (Infections and infestations) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiotoxicity (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 1
Ejection Fraction Decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TX05 (Trastuzumab) (N=394) | Herceptin® (N=400)
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 45 | 39
Peripheral Sensory Neuropathy (Nervous system disorders) | 33 | 30
Neuropathy Peripheral (Nervous system disorders) | 16 | 33
Nausea (Gastrointestinal disorders) | 27 | 31
Asthenia (General disorders) | 30 | 40
Alanine Aminotransferase Increased (Investigations) | 27 | 26
Aspartate Aminotransferase Increased (Investigations) | 19 | 12
Anemia (Blood and lymphatic system disorders) | 26 | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03556358/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT03556358/SAP_001.pdf